CLINICAL TRIAL: NCT05058573
Title: Effect of Temporomandibular Joint Disorder Relaxation and Myofacial Relaxation Techniques on Quality of Life, Depression and Headache in Individuals With Tension Headache
Brief Title: Effcet of Temporomandibular Joint Disorder Relaxation and Myofacial Relaxation Techniques on Tension Headache
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Ayça Araci, Physical Therapist,principal investigator, pHd, Alanya Alaaddin Keykubat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10354421-2021/07-08
Record Dates: First submitted 2021-09-09; First posted 2021-09-27 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Tension-Type Headache
Keywords: Tension - Type Headache; Temporomandibular Joint Disorder; Myofascial Release Techniques; Temporomandibular joint release techniques; Physiotherapy
MeSH Terms: conditions — Tension-Type Headache; Temporomandibular Joint Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Participant
Masking Description: it was calculated that 80% power could be achieved at a 95% confidence level when at least 66 people (at least 22 people for each group) were taken into the study. Therefore, our study Decocking TMJ+myofascial release+ a classic medical treatment (N= 25), TMJ Decocking+ classical medical treatment (N= 25), just the usual medical therapy (N=25) Group 3 group to be 75 individuals will be included. Assessments will be made before and after treatment. Treatment will be carried out in the form of 8 sessions in an average of 20-30 minute sessions 2 days a week for 4 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Myofascial relaxation technique + Temporomandibular joint release techniques group (n=22) (Experimental): medical treatment + temporomandibular joint relaxation (temporalis, masseter, and suboccipital muscles) + myofasial release/trigger points (trapezius, rhomboideus, and levator scapulae, sternocleidomastoideus muscles),
  Interventions: Other: Control group (n=22)
- Temporomandibular joint release techniques group (n=22) (Experimental): only temporomandibular joint relaxation will be performed in this group (temporalis, masseter, and suboccipital muscles).
  Interventions: Other: Control group (n=22)
- Control group (n=22) (Experimental): only medication treatment will be applied
  Interventions: Other: Control group (n=22)

INTERVENTIONS:
Other: Control group (n=22) — Control group will be received only medical treatment

SUMMARY:
The aim of this course is to investigate the effect of temporomandibular joint relaxation and myofacial relaxation techniques on quality of life , Joint range of motion, headache, depression in individuals with tension type headache.

DETAILED DESCRIPTION:
One of the most common complaints in society is headaches. Headaches affect the quality of life of people and communities.The proportion of people who have experienced headaches at least once in their lifetime is more than 90% in society, 93% in men and 99% in women.The causes that are common and cause this discomfort are basically examined under two main groups.These are grouped as 'primary/primary type headaches and secondary/secondary type headaches'. Some studies in literature have reported that temporomandibular dysfunction and headaches are 'comorbid diseases', that the presence of one will increase the symptoms of the other, and that if the temporomandibular joint disorder and headchache occur together, symptoms will shows sooner than expected.Some studies in literature have reported that temporomandibular dysfunction and headaches are 'comorbid diseases', that the presence of one will increase the symptoms of the other, and that if the temporomandibular joint disorder and the tension headaches occur together, it will show symptoms sooner than expected. The International Classification of Headache Disorders decodes the relationship between temporomandibular joint dysfunctions and headache.it is mentioned that as headache attributed to temporomandibular joint disorders. Many common points in studies have shown the Association of temporomandibular dysfunction and tension-type headache. The temporomandibular joint, one of the most complex joints in the body, is a loose joint that harmonizes between the mandibular condyle and the mandibular Fossa of the temporal bone decoction. The skull is the only movable joint between the bones decoction.November: the head and neck are a part of the stomatognathic system (masticatory system), which includes the muscles of the neck, chewing November, teeth-ligaments and salivary glands.Temporomandibular joint disorders are a major problem, covering approximately 5% to 12% of the population.Temporomandibular joint dysfunction leads to headaches, stiffness-pain in the jaw, restriction in jaw movements and stress increases TMD has been noted that the patients have difficulty doing daily life activities. Most Temporomandibular joint problems occur when the muscles around the joint are affected and pain occurs during the movements of the mandible and decreased functional use of the temporomandibular November. The muscles in the cervical region are also responsible for ensuring the stable position of the head, as well as for stabilizing the neck during movements of the jaw November. All November, the muscles in the craniocervical and facial region are connected. Temporomandibular joint dysfunctions (TMED) are more common in people with episodic tension headache (EGBTA) , migraine, and chronic tension headache (KGTBA) than in those without headache. When we look at literature, there are a limited number of studies in patients with Temporomandibular joint dysfunction with tension-type headache. Our study aimed to examine the effectiveness of temporomandibular joint relaxation and myofacial techniques on quality of life , Joint range of motion, headache, depression in individuals with tension type headache.

ELIGIBILITY:
Inclusion Criteria:

* individuals diagnosed with tension-type headache by a specialist physician
* individuals diagnosed with Temporomandibular joint dysfunction by dentist-maxillofacial surgeon
* To be able to read and understand Turkish
* Have not received any medical treatment in the last 1 year.

Exclusion Criteria:

* who received physical therapy for TMED in the previous 6 months
* who with any neurological problems
* who with any mental prolems
* who with any konjenital disorders
* who have undergone any cervikal or cranial surgery
* who have any facial trauma or facial paralyses
* who have advanced cervikal disc herniation
* who have ankylosing spondlitis, rhematoid arthritis, fibromyalgia
* who have any cominication problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-04-10 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-11-15 (Estimated)

PRIMARY OUTCOMES:
Cervikal region range of motion measurement | "baseline,preintervention " and "immediately after the intervention"
  Cases will be shown and asked to perform head flexion, extension, lateral flexion and rotation movements. And active joint range of motion will be evaluated with goniometer.
Temporomandibular joint range of motion measurement | "baseline,preintervention " and "immediately after the intervention"
  In our study, the maximum mouth opening amount of individuals in the group will be measured with a millimeter ruler 'right , left and side movements of the jaw (laterotrusion), forward movement (protrusion) and back movement (retrusion)'.
Fonseca Questionnare | "baseline,preintervention " and "immediately after the intervention"
  In order to classify Temporomandibular joint dysfunction, the Fonseca questionnaire will be applied. this questionnaire consists of 10 questions. Participants are asked to answer each question in the form of Yes (10 points), Sometimes (5 points ), No (0 points). Scores of all questions are collected and the severity of temporomandibular joint dysfunction is determined. TMED-No (0-15 points), Mild-TMED (20-40 points), Moderate-TMED (45-60 points) and Severe - TMED (70-100 points).
Headache Impact Test | "baseline,preintervention " and "immediately after the intervention"
  This questionnaire describes the frequency of a person's headache, the degree of restriction in daily life activities and social settings due to headaches , their psychological state , changes in their cognitive function.
Beck depression scale | "baseline,preintervention " and "immediately after the intervention"
  In order to evaluate depression level, The beck depression scale will be used.in the scale consisting of 21 questions, each question consists of 4 styles. The questions are scored between 0-3 points dec Low scores represent good results. According to the scores obtained, (0-9) points indicate minimal depression, (10-16) points indicate mild depression, (17-29) points indicate moderate depression, and (30-63) points indicate severe depression
Beck Anxiety Sacle | "baseline,preintervention " and "immediately after the intervention"
  In order to evaluate anxiety level, The beck depression scale will be used.in this scale consisting of 21 items, a quadruple Likert type measurement is performed. 0 points = none ,1 point = light , 2 points =medium , 3 points = serious. the december of 8-15 points is expressed as mild anxiety symptoms, moderate anxiety dec 16-25 points, severe anxiety symptoms from 26-63 points.
General short form quality of life scale | "baseline,preintervention " and "immediately after the intervention"
  In order to evaluate the quality of life, the short form quality of life will be used.SF-36 is a test consisting of 36 items used to obtain information about a person's physical, emotional, and general health status. This test includes 8 subscales ; mental state ,energy, pain, physical function, limitation due to physical problems, restriction due to emotional problems, social function and general health. it is evaluated with a score of 0-100 points.dec. High marks indicate a good state of health.

CONTACTS AND LOCATIONS:
Overall Officials: Hanifegül Taşkıran, Prof. Dr, Study Chair — İstanbul Aydın University; Mustafa Zafer DEMİRTAŞ, MD, Study Director — Alanya Alaaddin Keykubat University; Ertan KARAÇAY, MD, Study Director — Alanya Alaaddin Keykubat University; Ahmet ÖZŞİMŞEK, PHD MD, Study Director — Alanya Alaaddin Keykubat University
Locations (1):
- Alanyaaku, Antalya, Alanya, Turkey (Türkiye)